CLINICAL TRIAL: NCT00384514
Title: A Study for Testing Safety and Efficacy of the Administration of Blood-Borne Autologous Endothelial Progenitor Cells to Alleviate Anginal Symptoms and Myocardial Ischemia in Patients With Severe Anginal Syndrome
Brief Title: EPC by Intracoronary Injection in Patients With Chronic Stable Angina
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TheraVitae Ltd. (Industry)
Collaborators: Mahidol University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TV-001
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2006-10-20 (Estimated); Status verified 2006-10

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery disease with chronic stable angina
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Device: VesCell (TM)-Autologous EPCs/Angiogenic Cell Precursors

SUMMARY:
Study title:A Study for Testing Safety and Efficacy of the administration of Blood-Borne Autologous Endothelial Progenitor Cells to Alleviate Anginal Symptoms and Myocardial Ischemia in Patients with Severe Anginal Syndrome

Principle Investigator: Assoc. Prof. Damras,Tresukosol,M.D.,Head of Cardiac Catherlization unit,Division of Cardiology,Department of Medicine,Faculty of Medicine Siriraj Hospital,Mahidol University

Study objective : To determine the safety and efficacy of intracoronary injection of blood-borne autologous EPCs in relieving symptoms of angina pectoris in symptomatic patients treated with maximal medical therapy with an occluded coronary artery supplying ischemic myocardium Study Design : Phase II, a single center,a non-randomized,open-label trial,

Study population :

Total expected no. of patients : 24

main selection criteria :

* Patients with chronic stable angina on maximal medical therapy and an occluded coronary artery supplying an ischemic viable myocardial region as shown on Sesta-mibi scan. On coronary angiography,the occluded coronary artery must have a patent proximal segment of at least 30 mm with at least one side branch to enable the injection of the EPC if the vessel remains occluded despite the attempted angioplasty efforts.
* Age 18-80 years
* Ejection fraction >35 % on Sesta-mibi scan
* Sestamibi scan (myocardial perfusion) during exercise or dipyridamole,demonstrating regional reversible ischemia in an area relating to the occluded coronary artery.

Investigational Product : At D-8 250 ml of blood drawn from the patients for production of autologous EPCs or ACPs (VescellTM), On D0 ,at least 1.5 million EPCs with viability >75 % suspended in 6 ml sterile cell culture medium will be injected to the same patients by intracoronary artery.

The study consists of 4 periods:Screening ( D-14to-9&D-8,Treatment(D0),Acute Safety follow-up (D1&D2),Chronic follow-up (D30,D90&D180)period ,total follow-up of each case is 6 months.

Evaluation criteria :

Safety : no.& duration of adverse event & serious adverse event

Efficacy :

* change from baseline to 1,3,6 months of CCS, 6-minute walking test
* change from baseline to 3 & 6 months of Sesta-mibi scan
* change from baseline to 3 & 6 months of symptom-limited exercise time,exercise-induced ischemia & METs on Sesta-mibi scan Duration of study: July 2004-December 2006

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic stable angina on maximal medical therapy and an occluded coronary artery supplying an ischemic viable myocardial region as shown on Sestamibi scan. On coronary angiography, the occluded coronary artery must have a patent proximal segment of at least 30 mm with at least one side branch to enable the injection of the EPC if the vessel remains occluded despite the attempted angioplasty efforts.
* Patients are not candidates for or are not willing to undergo CABG surgery.
* Age 18 to 80 years
* Male or non-pregnant, non-lactating female
* Ejection fraction >35% on Sestamibi
* Sestamibi scan (myocardial perfusion) during exercise or dipyridamole, demonstrating regional reversible ischemia in an area relating to the occluded coronary artery.
* Informed consent obtained and consent form signed

Exclusion Criteria:

* Patients not satisfying the coronary angiography and Sestamibi criteria
* Patient who received blood transfusions during the previous 4 weeks (to exclude the potential of non-autologous EPCs in the harvested blood).
* Inability to communicate (that may interfere with the clinical evaluation
* Myocardial infarction during the preceding 3 months
* Significant valvular disease or after valve replacement
* After heart transplantation
* Cardiomyopathy
* Renal failure (creatinine 10% above the upper limit according to the hospital normograms)
* Hepatic failure
* Anemia (lower than 11mg/dl.hemoglobin for female and lower than 12 mg/dl for male)
* Abnormal coagulation tests normal [platelets, PT (INR), PTT]
* Stroke within the preceding 3 years
* Malignancy within the preceding 3 years
* Concurrent chronic or acute infectious disease
* Severe concurrent medical disease (e.g., septicemia, HIV-1,2/HBV/HCV infections, insulin-dependent diabetes mellitus, systemic lupus erythematosus, multiple sclerosis, amyotrophic lateral sclerosis)
* Chronic immunomodulating or cytotoxic drugs treatment
* Patients who have rectal temp. above 38.40C for 2 consecutive days
* Patient unlikely to be available for follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2004-07; Study Completion 2006-09

PRIMARY OUTCOMES:
Safety : no.& duration of adverse event & serious adverse event
Efficacy :change from baseline to 1,3,6 months of CCS, 6-minute walking test

SECONDARY OUTCOMES:
Efficacy : change from baseline to 3 & 6 months of Sesta-mibi scan
: change from baseline to 3 & 6 months of symptom-limited exercise time,exercise-induced ischemia & METs on Sesta-mibi scan

CONTACTS AND LOCATIONS:
Overall Officials: Damras Tresukosol, M.D., Principal Investigator — Head of Cardiac Catherlization unit,Division of Cardiology,Department of Medicine,Faculty of Medicine Siriraj Hospital,Mahidol University ,BKK,Thailand
Locations (1):
- Dr. Valentin Fulga, Kiryat Weizmann Science Park, Nes Zionna, Israel